CLINICAL TRIAL: NCT06131060
Title: Effects of Progressive Eccentric Exercises Verses Bodyweight Exercises on Agility, Power and Functional Performance in Athletes With Hamstring Strain.
Brief Title: Progressive Eccentric VS Bodyweight Exercises on Agility, Power and Functional Performance in Hamstring Strain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0443
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Exercise Movement Techniques; Exercise Therapy; Hamstring Injury
Keywords: Progressive eccentric exercises; Bodyweight exercises; Hamstring strain

STUDY DESIGN:
Intervention Model Description: Randomized clinical trials
Who Masked: Outcomes Assessor
Masking Description: The assessor who will take the readings is blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive eccentric exercises (Experimental): Group A will perform progressive eccentric exercises that includes eccentric squats, Nordic hamstring curls and reverse Nordic hamstring curls.
  Three sessions per week for 6 weeks.
  Interventions: Other: Progressive eccentric exercises
- Bodyweight exercises (Experimental): Group B will perform bodyweight exercises that includes Bulgarian split squat, Glut-Ham bridge, sliding leg curl.
  Three sessions per week for 6 weeks.
  Interventions: Other: Bodyweight exercises

INTERVENTIONS:
Other: Progressive eccentric exercises — This include progressive eccentric exercises thrice a week for 6 weeks.
  Arms: Progressive eccentric exercises
Other: Bodyweight exercises — This include bodyweight exercises thrice a week for 6 weeks
  Arms: Bodyweight exercises

SUMMARY:
The study is randomized and single blinded. Ethical approval is taken from ethical committee of Riphah international university Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A and group B through sealed envelope method by non probability convenient random sampling technique. Subjects in group A will receive Progressive eccentric exercises. Group B will receive Bodyweight exercises.

DETAILED DESCRIPTION:
The objective of the study is to determine the effects of progressive eccentric exercises verses Bodyweight exercises on agility, power and functional performance in athletes with hamstring strain. The study is randomized and single blinded. Ethical approval is taken from ethical committee of Riphah international university Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A and group B through sealed envelope method by non probability convenient random sampling technique. Subjects in group A will receive Progressive eccentric exercises. Group B will receive Bodyweight exercises. The outcome measures will be assessed by T test, Vertical jump, Standing Long jump and squat test. The data will be analyzed by SPSS, Version 25. Statistical significance is P=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Athletes older than of 18 years will be added. Athletes having history of Hamstring Strain of Grade 1 and 2.Participants will be added after 4 weeks of recovery period after grade 1 & 2 hamstring Strain.Male and female Athletes will be added.

Exclusion Criteria:

* Athletes with a complete rupture of the hamstring muscle. Athletes undergone hamstring surgery in the past 6 months will not be considered.Participants with history of back pain.Lower limb injuries in past 6 months.

If the hamstring strain is accompanied by severe associated injuries, such as fracture or significant ligament tear.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Agility | Pre and 6 weeks post interventional.
  Agility will be measured by T test.
Power | Pre and 6 weeks post interventional
  Power will be measured by vertical jump test and standing long jump test.
Functional performance | Pre and 6 weeks post interventional
  Functional performance will be measured by squat test

CONTACTS AND LOCATIONS:
Overall Officials: Raafia, DPT, Principal Investigator — Study principal investigator
Locations (1):
- Alfateh sports complex, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Horst N, Smits DW, Petersen J, Goedhart EA, Backx FJ. The preventive effect of the nordic hamstring exercise on hamstring injuries in amateur soccer players: a randomized controlled trial. Am J Sports Med. 2015 Jun;43(6):1316-23. doi: 10.1177/0363546515574057. Epub 2015 Mar 20. PMID 25794868
- [Background] Yoon SY, Kim YW, Shin IS, Kang S, Moon HI, Lee SC. The Beneficial Effects of Eccentric Exercise in the Management of Lateral Elbow Tendinopathy: A Systematic Review and Meta-Analysis. J Clin Med. 2021 Sep 1;10(17):3968. doi: 10.3390/jcm10173968. PMID 34501416
- [Background] Croisier JL, Forthomme B, Namurois MH, Vanderthommen M, Crielaard JM. Hamstring muscle strain recurrence and strength performance disorders. Am J Sports Med. 2002 Mar-Apr;30(2):199-203. doi: 10.1177/03635465020300020901. PMID 11912088
- [Background] Anderson CE, Sforzo GA, Sigg JA. The effects of combining elastic and free weight resistance on strength and power in athletes. J Strength Cond Res. 2008 Mar;22(2):567-74. doi: 10.1519/JSC.0b013e3181634d1e. PMID 18550975
- [Background] Maclachlan L, White SG, Reid D. OBSERVER RATING VERSUS THREE-DIMENSIONAL MOTION ANALYSIS OF LOWER EXTREMITY KINEMATICS DURING FUNCTIONAL SCREENING TESTS: A SYSTEMATIC REVIEW. Int J Sports Phys Ther. 2015 Aug;10(4):482-92. PMID 26346642